Official Title: A Phase IIa, Multicenter, Randomized, Placebo-Controlled, Double-

Blind Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of

MTPS9579A in Patients with Asthma Requiring Inhaled

Corticosteroids and a Second Controller

NCT Number: NCT04092582

**Document Date:** DAP Version 3: 30-July-2022

### **Output Specifications**

| Study title: | A PHASE IIA, MULTICENTER, RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND STUDY TO EVALUATE THE EFFICACY, SAFETY, AND PHARMACOKINETICS OF MTPS9579A IN PATIENTS WITH ASTHMA REQUIRING INHALED CORTICOSTEROIDS AND A SECOND CONTROLLER | |
|---|---|---|
| Protocol number: | GB41149 | |
| Reporting event: | CSR, August 2022 | |
| Author: | | |
| | | July 21,<br>2022 |
| Study Statistician | | Date |
| Approver: | | |
| | | July 30, 2022 |
| | | Date |

\* The approver has ensured that key team members have been involved, contributed, and reviewed the Output Specifications for completeness and ability to address the scientific objectives and reporting needs, as well as for appropriate level of scope.

### **Key Definitions:**

#### **Analysis Populations**

#### Intent-to-Treat (ITT) Population:

Definition: All patients who are randomized in the study.

Variable: ADSL.ITFL

#### Modified Intent-to-Treat (mITT) Population:

Definition: All patients randomized who received at least one dose of study drug.

Variable: ADSL.MITTFL

#### Run-in Safety-Evaluable (PEFL) Population:

Definition: All patients who received the single-blind placebo dose during the run-in period, regardless

of whether or not the patient is randomly allocated into the double-blind treatment period.

Variable: ADSL.PEFL

#### Safety-Evaluable (SE) Population:

Definition: All randomized patients who received at least one dose of study drug during the 48-week double-blind treatment period, with patients grouped according to treatment received (MTPS9579A or placebo)

Variable: ADSL.SAFFL

#### Biomarker Subgroups

- NASO
- SERUM

#### **Definition of Baseline**

Use randomization (Week 2) as the baseline.

- ADLB uses VISIT = "WEEK 2-RANDOMIZATION" for Baseline calculations; use VISIT = "SCREENING" for parameters that don't have VISIT = "WEEK 2-RANDOMIZATION".
- ADVS uses VISIT = "WEEK 2-RANDOMIZATION" and VSTPT = "PRE-DOSE" for Baseline calculations or VISIT = "SCREENING" for parameters that don't have VISIT = "WEEK 2-RANDOMIZATION" (height and weight).

### Data Handling Specifications:

General Output Specification Categories for all TLGs unless specified below:

Column Variables:

All outputs are unblinded. Columns are displayed in this order: 'Placebo', 'MTPS9579A'.

- Treatment Group: Group by Treatment Assigned. ADSL.TRT01P
- Column Totals: 'All Patients'
- Analysis Variables: See each mock-up below.
- **Numeric Precision and Formatting of Statistics**: Round to 1 decimal unless otherwise specified. For change from baseline outputs, using default STREAM precision is fine.
- Optional Subsetting: N

### Section 1. Study Conduct and Analysis Population

### **Output 1.1 Summary of Analysis Populations (APT01)**

Analysis Populations, Placebo Run-in Period, All Patients Protocol: GB41149

| | All Patients<br>(N=140) |
|-------------------------------------------|-------------------------|
| Run-in Safety-Evaluable (PEFL) Population | 140 ( 100%) |

Analysis Populations, All Patients

Protocol: GB41149

| | Placebo<br>(N=66) | MTPS9579A Active<br>(N=69) | All Patients<br>(N=135) |
|---|---|---|---|
| Intent-to-Treat Population (as Randomized) | 66 (100%) | 69 (100%) | 135 ( 100%) |
| Modified Intent-to-Treat Population | 65 (98.5%) | 69 (100%) | 134 (99.3%) |
| Safety-Evaluable Population | 65 (98.5%) | 69 (100%) | 134 (99.3%) |

### Output 1.2 Enrollment by Country and Investigator Number (ENT01A)

Protocol: GB41149

| Country,<br>Investigator Number | Placebo<br>(N=nnn) | MTPS9579A<br>(N=nnn) | All Patients<br>(N=nnn) |
|---|---|---|---|
| Country 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Country 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Country 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### **Output 1.3 Summary of Major Protocol Deviations (PDT01)**

Protocol: GB41149

Analysis Population: Intent-to-treat population

| Category | Placebo | MTPS9579A | All Patients |
|---|---|---|---|
| Description | (N=nnn) | (N=nnn) | (N=nnn) |
| Total number of patients with at least one major protocol deviation | nn(xx.x%) | nn (xx.x%) | nn(xx.x%) |
| Total number of major protocol deviations | nn | nn | nn |
| Inclusion Criteria | | | |
| Number of patients | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Exclusion Criteria | | | |
| Number of patients | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Procedural deviation | | | |

### **Output 1.4 Listing of Major Protocol Deviations (PDL01)**

Protocol: GB41149

Analysis Population: Intent-to-treat population

Treatment: PLACEBO

| Subject Identifier | Major | Deviation |
|---|---|---|
| | Yes<br>Yes<br>Yes | Inclusion criteria<br>Exclusion criteria<br>Procedural |

### **Output 1.5 Patient Disposition (DST01)**

Protocol: GB41149

| Status | Placebo<br>(N=nnn) | MTPS9579A<br>(N=nnn) | All Patients<br>(N=nnn) |
|---|---|---|---|
| Completed study | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Optional row 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Optional row 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Optional row n | | | |
| Discontinued study | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Reason 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Reason 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### Output 1.6 Patients Discontinued from Study Treatment (DST01)

Protocol: GB41149

| Status | Placebo<br>(N=nnn) | MTPS9579A<br>(N=nnn) | All Patients<br>(N=nnn) |
|---|---|---|---|
| Completed treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Optional row 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Optional row 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Optional row n | | | |

| Discontinued treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
|------------------------|------------|------------|------------|
| Reason 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Reason 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### Output 1.7 Listing of Patients who Discontinued from Study (DSL02)

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population

Treatment: PLACEBO

| Center/<br>Patient ID | \ge/Sex/Race | Date of First<br>Study Drug<br>Administration | ay of Last Study<br>Drug<br>Administration | Day of Study<br>Discontinuation<br>Relative to First<br>Study Drug<br>Administration | Day of Study<br>Discontinuation<br>Relative to<br>Randomization | leason for Discontinuation |
|---|---|---|---|---|---|---|
| | /Fi | | 12 | 14 | 14 | Adverse event |
| | /M/ | | 36 | 65 | 65 | Lost to follow-up |
| | /Ma | | | | 2 | Withdrawal by subject |

# Output 1.8 Listing of Patients who Discontinued from Study Treatment (DSL02)

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population

Treatment: PLACEBO

| Center/<br>Patient ID | Age/<br>Sex/Race | Date of First<br>Study Drug<br>Administration | Day of Last<br>Study Drug<br>Administration | Day of Treatment<br>Discontinuation<br>Relative to First<br>Study Drug<br>Administration | Day of Treatment<br>Discontinuation<br>Relative to<br>Randomization | Reason for<br>Discontinuation |
|---|---|---|---|---|---|---|
| | /F/ | | 12 | 14 | 14 | Adverse event |
| | /M/ | | 36 | 65 | 65 | Lost to follow-up |
| | /M | | | | 2 | Withdrawal by subject |

### Section 2 Demographics & Baseline Characteristics

### Output 2.1 Demographics and Baseline Characteristics (DMT01)

Protocol: GB41149

| | Placebo<br>(N = XXX) | MTPS9579A<br>Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|
| Age (yr) | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | xx.x |
| Min-max | XX-XX | xx-xx | XX-XX |
| Age group (yr) | | | |

| n | nnn | nnn | nnn |
|---------------------------|------------|------------|------------|
| 18 – <50 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 50 – <65 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >= 65 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Sex | | | |
| n | nnn | nnn | nnn |
| Male | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Female | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Ethnicity | | | |
| n | nnn | nnn | nnn |
| Hispanic or Latino | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Not Hispanic or Latino | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Race | | | |
| n | nnn | nnn | nnn |
| Asian | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Black or African American | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

| White | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
|-------------------------|-------------|-------------|-------------|
| Unknown | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Weight (kg) at Baseline | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x | Xx.x- |
| Min-max | xx.x | xx.x | xx.x |
| Height (cm) at Baseline | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x | xx.x |
| Min-max | xx.x | xx.x | xx.x |
| BMI (kg/m2) at Baseline | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x | XX.X |

| Min-max | XX.X | xx.x | xx.x |
|---|---|---|---|
| Geographic Region, IxRS Stratif | | | |
| n | nnn | nnn | nnn |
| United States / Western Europe | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Eastern Europe | XX.X | xx.x | xx.x |
| Southern Hemisphere | XX.X | xx.x | xx.x |
| Asthma Exac in Prior Year, IxRS Stratif | | | |
| n | nnn | nnn | nnn |
| 1 event | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| >=2 events | XX.X | xx.x | xx.x |
| Percent Predicted FEV1 at Baseline | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x | xx.x |
| Min-max | XX.X | xx.x | xx.x |
| Blood Eosinophils at Baseline | | | |

| n | nnn | nnn | nnn |
|---|---|---|---|
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x | XX.X |
| Min-max | xx.x | xx.x | xx.x |
| Blood Eosinophils Group at Baseline | | | |
| n | nnn | nnn | nnn |
| < 150 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 150 - 300 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| > 300 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Active Tryptase Allele Counts | | | |
| n | nnn | nnn | nnn |
| <=2 | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| >2 | xx.x | xx.x | xx.x |
| ACQ-5 Score at Baseline | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |

| Median | XX.X | XX.X | XX.X |
|---------|-------|-------|-------|
| Min-max | xx-xx | xx-xx | xx-xx |

### Output 2.2 Listing of Investigators (ENL01)

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population

| Center | Investigator | Investigator Number | Center Name | Country |
|--------|--------------|---------------------|-------------|---------|

### Output 2.3 Listing of Demographics and Baseline Characteristics (DML01)

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population

Treatment: <Treatment>



### Output 2.4 Listing of Randomization Assignments (DML02)

Protocol: GB41149

| Center/Patient ID | Randomized | Date of | Date of |
|---|---|---|---|
| | Treatment | Randomization | First Study Drug Administration |
| | | | Administration |



Placebo
Placebo
Placebo
Active Treatment
Active Treatment
Active Treatment
Active Treatment





### **Output 2.5 Summary of Medical History (MHT01)**

Protocol: GB41149

Analysis Population: Run-in safety-evaluable population (PEFL)

| MedDRA System Organ Class<br>MedDRA Preferred Term | Placebo<br>(N = XXX) | MTPS9579A<br>(N = XXX) | All Patients<br>(N=nnn) |
|---|---|---|---|
| Total number of patients with at least one condition | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of conditions | nnn | nnn | nnn |
| VASCULAR DISORDERS | | | |
| Total number of patients with at least one condition | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of conditions | nn | nn | nn |
| HYPERTENSION | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| VARICOSE VEINS | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Investigator text for medical history conditions coded using MedDRA version xx.x. Percentages are based on N in the column headings.

Includes all diseases and conditions reported as part of asthma medical history, categorized by Clinical Science.

### **Output 2.6 Listing of Medical History (MHL01)**

Protocol: GB41149

Analysis Population: Run-in safety-evaluable population (PEFL)

Treatment: ARM A



Investigator text for medical history conditions coded using MedDRA xx.x.

### Output 2.7 Glossary of Medical History Coded Terms (AEL01\_NOLLT)

Protocol: GB41149

Analysis Population: Run-in safety-evaluable population (PEFL)

| MedDRA System Organ Class Specified Medical History Term | MedDRA Preferred Term | Investigator- |
|---|---|---|
| BLOOD AND LYMPHATIC SYSTEM DISORDERS<br>DEFICIENCY ANAEMIA | IRON DEFICIENCY ANAEMIA | IRON |
| CONGENITAL, FAMILIAL AND GENETIC DISORDERS | ARNOLD-CHIARI MALFORMATION | ARNOLD |
| CHIARI | GILBERT'S SYNDROME | GILBERT'S |
| SYNDROME | | |

<sup>\*</sup> End day derived from imputed end date.

...

### Section 3. Efficacy Analysis

Efficacy analyses will be conducted on an mITT population, consisting of all randomized patients who received at least one dose of study drug during the 48-week double-blind treatment period, with patients grouped according to the treatment assigned at randomization.

Unless otherwise noted, analyses of efficacy outcome measures will be adjusted by:

- 1. Blood eosinophil level at week 2 randomization visit (<u>ADSL.BEOGRWK2</u> < 150 cells/ $\mu$ L, 150-300 cells/ $\mu$ L, > 300 cells/ $\mu$ L)
- 2. Geographic region (<u>ADSL.REGIONST</u>: United States/Western Europe, Eastern Europe, Southern Hemisphere)
- 3. Asthma exacerbations in prior year (ADSL.ASMEXGST)

#### **Tables**

### Output 3.1 Time to First CompEx Event, 48-Week Double-Blind Treatment Period

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (MITTFL = 'Y')

| | Placebo | MTPS9579A Active |
|-----------------------------------|------------|------------------|
| Total number of patients per arm | XX | XX |
| Patients with event: N (%) | XX (XX.X%) | XX (XX.X%) |
| Patients with diary event: N (%) | XX (XX.X%) | XX (XX.X%) |
| Patients with exacerbation: N (%) | XX (XX.X%) | XX (XX.X%) |
| Patients without event (%) | XX (XX.X%) | XX (XX.X%) |

| Median | XXX.X | XXX.X |
|---------------------|------------|--------------|
| 95% CI | (XXX, XXX) | (XXX, XXX) |
| 25 - 75 percentile | XXX, XXX | XXX, XXX |
| Range | XXX to XXX | XXX to XXX |
| Stratified Analysis | | |
| p-value (log-rank) | - | X.XXXX |
| Hazard Ratio | - | x.xx |
| 95% CI | - | (XX.X, XX.X) |
| p-value | - | X.XXXX |

Hazard ratios were estimated by Cox regression with the following stratification factors as covariates: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region (United States/Western Europe [United States, Germany], Eastern Europe [Poland], Southern Hemisphere [Peru, Argentina]).

## Output 3.2 Time to First Protocol-Defined Asthma Exacerbation, 48-Week Double-Blind Treatment Period

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (MITTFL = 'Y')

| Time to First Protocol-defined Asthma Exacerbation, 48–Week Double–Blind Treatment Period, mITT Subjects Who Were Dosed in Treatment Period | | |
|---|---|---|
| | Placebo | MTPS9579A Active |
| Total number of patients per arm | XX | XX |
| Patients with event (%) | XX (XX.X%) | XX (XX.X%) |
| Patients without event (%) | XX (XX.X%) | XX (XX.X%) |
| Time to event (weeks) | | |
| Median | XXX.X | XXX.X |
| 95% CI | (XXX, XXX) | (XXX, XXX) |

| 25 - 75 percentile | XXX, XXX | XXX, XXX |
|---------------------|------------|--------------|
| Range | XXX to XXX | XXX to XXX |
| Stratified Analysis | | |
| p-value (log-rank) | - | X.XXXX |
| Hazard Ratio | - | X.XX |
| 95% CI | - | (XX.X, XX.X) |
| p-value | - | X.XXXX |

Hazard ratios were estimated by Cox regression with the following stratification factors as covariates: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region (United States/Western Europe [United States, Germany], Eastern Europe [Poland], Southern Hemisphere [Peru, Argentina]).

## Output 3.3 Rate of Asthma Exacerbations, 48-Week Double-Blind Treatment Period

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (MITTFL = 'Y')

Rate of Protocol-defined Asthma Exacerbation, 48-Week Double-Blind Treatment Period, All mITT Subjects Who Were Dosed in Treatment Period

| | Placebo | MTPS9579A Active |
|-------------------------------------|------------|------------------|
| N | XXX | XXX |
| Number of exacerbations per patient | | |
| 0 | XX (XX.X%) | XX (XX.X%) |
| 1 | XX (XX.X%) | XX (XX.X%) |
| 2 | XX (XX.X%) | XX (XX.X%) |
| 3 | XX (XX.X%) | XX (XX.X%) |
| Total number of exacerbations | XXX | XXX |

| Total follow-up time at risk (years) | XXX.X | XXX.X |
|---|---|---|
| Exacerbation rate (per year) | | |
| Unadjusted | X.XX | X.XX |
| Adjusted | X.XX | X.XX |
| Absolute rate difference (events/ year), adjusted (MTPS9579A - placebo) | _ | X.XX |
| Rate ratio, adjusted (MTPS9579A/placebo) | _ | X.XX |
| 95% CI | | (X.XX, X.XX) |
| p-value | _ | X.XXXX |
| Percentage rate reduction, adjusted (MTPS9579A vs. placebo) | _ | (XX.X%) |

Adjusted exacerbation rates and rate ratio are estimated from a Poisson regression model with over-dispersion adjusted for the following covariates and log(patient time at risk) as offset term: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region (United States/Western Europe [United States, Germany], Eastern Europe [Poland], Southern Hemisphere [Peru, Argentina]).

# Output 3.4 Pre-Bronchodilator FEV1 Results and Change from Baseline by Visit (L), 48-Week Double-Blind Treatment Period

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FEV1 MITT = 'Y')

| | | | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) |
|---|---|---|---|---|
| Baseline Value at vis | Value at visit | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |

| Week 3 | Value at visit | n | XXX | XXX |
|---|---|---|---|---|
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Change from baseline | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Percent change from | _ | XXX | VVV |
| | baseline | n<br>Mean (SD) | XX.X (XX.X) | XXX<br>XX.X (XX.X) |
| | | Median | XX.X (XX.X) | XX.X (XX.X) |
| | | Min - Max | XX.X (XX.X) | XX.X (XX.X) |
| Week | | | | |
| Week 50 | Value at visit | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Change from baseline | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | xxxx |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Percent change from baseline | n | XXX | XXX |
| | | Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |

| Median | XX.X (XX.X) | XX.X (XX.X) |
|-----------|-------------|-------------|
| Min - Max | XX.X (XX.X) | XX.X (XX.X) |

# Output 3.5 Pre-Bronchodilator FeNO Results and Change from Baseline by Visit (ppb), 48-Week Double-Blind Treatment Period

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FENO\_MITT = 'Y')

Pre-Bronchodilator FeNO Results and Change from Baseline by Visit (ppb), 48–Week Double-Blind Treatment Period, mITT Subjects Who Were Dosed in Treatment Period

| | | | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) |
|---|---|---|---|---|
| Baseline | Value at visit | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| Week 3 | Value at visit | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Change from baseline | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Percent change from baseline | n | XXX | XXX |
| | | Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |
| | | Median | XX.X (XX.X) | XX.X (XX.X) |
| | | Min - Max | XX.X (XX.X) | XX.X (XX.X) |

| Week | | | | |
|---|---|---|---|---|
| vveek | | | | |
| Week 50 | Value at visit | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | xxxx |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Change from baseline | n | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) |
| | | Median | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX |
| | Percent change from baseline | n | XXX | XXX |
| | | Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |
| | | Median | XX.X (XX.X) | XX.X (XX.X) |
| | | Min - Max | XX.X (XX.X) | XX.X (XX.X) |

# Output 3.6 Mixed-Effect Model Repeated Measures Analysis of <u>Absolute</u> Change from Randomization Visit in Pre-bronchodilator FEV1 (L) through Week 50

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FEV1\_MITT = 'Y')

Mixed-Effect Model Repeated Measures Analysis of Absolute Change from Randomization Visit in Pre-bronchodilator FEV1 (L) through Week 50, mITT Subjects Who Were Dosed in Treatment Period

| Visit | Absolute Change from Baseline, Pre-Bronchodilator FEV1 (L) | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) |
|---|---|---|---|
| Week 3 | n | XXX | XXX |
| | Adjusted Mean (SE) | XXX (XX) | XXX (XX) |
| | 95% CI for Adjusted Mean | (XXX, XXX) | (XXX, XXX) |
| | Difference in Adjusted Means (SE) | - | XXX (XX) |

| | 95% CI for Difference in Adjusted Means | - | (XXX, XXX) |
|---------|-----------------------------------------|------------|------------|
| | P-value | - | X.XXXX |
| Week | | | |
| Week 50 | n | XXX | XXX |
| | Adjusted Mean (SE) | XXX (XX) | XXX (XX) |
| | 95% CI for Adjusted Mean | (XXX, XXX) | (XXX, XXX) |
| | Difference in Adjusted Means (SE) | - | XXX (XX) |
| | 95% CI for Difference in Adjusted Means | - | (XXX, XXX) |
| | P-value | - | X.XXXX |

Footnotes: Estimates are based on a mixed model for repeated measures (MMRM) analysis with an unstructured covariance matrix. The model used the absolute change pre-bronchodilator FEV1 as the response variable and included terms for treatment arm, study visit, treatment arm by study visit interaction, baseline FEV1 as well as its interaction with study visit, in addition to the stratification factors: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region (United States/Western Europe [United States, Germany], Eastern Europe [Poland], Southern Hemisphere [Peru, Argentina]). Subjects without valid baseline values are excluded from analysis.

N in the header represents the number of subjects with at least one post-baseline value.

# Output 3.7 Mixed-Effect Model Repeated Measures Analysis of <u>Relative</u> Change from Randomization Visit in Pre-bronchodilator FEV1 (L) through Week 50

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FEV1 MITT = 'Y')

Similar to Output 3.6.

# Output 3.8 Mixed-Effect Model Repeated Measures Analysis of <u>Absolute</u> Change from Randomization Visit in FeNO (ppb) through Week 50

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FENO MITT = 'Y')

Mixed-Effect Model Repeated Measures Analysis of Absolute Change from Randomization Visit in Pre-bronchodilator FeNO (ppb) through Week 50, mITT Subjects Who Were Dosed in Treatment Period

| Visit | Absolute Change from Baseline,<br>Pre-Bronchodilator FeNO (ppb) | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) |
|---|---|---|---|
| Week 3 | n | XXX | XXX |
| | Adjusted Mean (SE) | XXX (XX) | XXX (XX) |
| | 95% CI for Adjusted Mean | (XXX, XXX) | (XXX, XXX) |
| | Difference in Adjusted Means (SE) | - | XXX (XX) |
| | 95% CI for Difference in Adjusted Means | - | (XXX, XXX) |
| | P-value | - | X.XXXX |
| Week | | | |
| Week 50 | n | XXX | XXX |
| | Adjusted Mean (SE) | XXX (XX) | XXX (XX) |
| | 95% CI for Adjusted Mean | (XXX, XXX) | (XXX, XXX) |
| | Difference in Adjusted Means (SE) | - | XXX (XX) |
| | 95% CI for Difference in Adjusted Means | - | (XXX, XXX) |
| | P-value | - | X.XXXX |

Footnotes: Estimates are based on a mixed model for repeated measures (MMRM) analysis with an unstructured covariance matrix. The model used the absolute change pre-bronchodilator FeNO as the response variable and included terms for treatment arm, study visit, treatment arm by study visit interaction, baseline FeNO as well as its interaction with study visit, in addition to the stratification factors: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region (United States/Western Europe [United States, Germany], Eastern Europe [Poland], Southern Hemisphere [Peru, Argentina]).

N in the header represents the number of subjects with at least one post-baseline value.

# Output 3.8 Mixed-Effect Model Repeated Measures Analysis of Relative Change from Randomization Visit in FeNO (ppb) through Week 50

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FENO MITT = 'Y')

Similar to Output 3.7.

### Graphs

## Output 3.9 Time to First CompEx Event, 48-Week Double-Blind Treatment Period

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (MITTFL = 'Y')

Kaplan Meier Plot of Time to First CompEx Event, 48-Week Double-Blind Treatment Period, mITT Subjects Who Were Dosed in Treatment Period

## Output 3.10 Time to First Protocol-Defined Asthma Exacerbation, 48-Week Double-Blind Treatment Period

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (MITTFL = 'Y')

Kaplan Meier Plot of Time to First Protocol-defined Asthma Exacerbation, 48-Week Double-Blind Treatment Period, mITT Subjects Who Were Dosed in Treatment Period

# Output 3.11 Absolute Change from Randomization in Pre-bronchodilator FEV1 (L) Across Time

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FEV1 MITT)

Note: add the number of patients at each time point in the plot. Considering the applicability of SAS, a separate table placed below the plot is also acceptable.

# Output 3.12 Relative Change from Randomization in Pre-bronchodilator FEV1 (%) Across Time

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FENO\_MITT)

Similar to Output 3.11.

# Output 3.13 Absolute Change from Randomization in Pre-bronchodilator FeNO (ppb) Across Time

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FENO\_MITT)

Similar to Output 3.11.

# Output 3.14 Relative Change from Randomization in Pre-bronchodilator FeNO (%) Across Time

Protocol: GB41149

Analysis Population: Modified Intent-to-treat population (FEV1\_MITT)

Similar to Output 3.11.

### Section 4. Safety Analysis

#### **Tables**

#### **Output 4.1 Study Treatment Exposure (EXT01)**

Protocol: GB41149

Analysis Population: Double-Blind Treatment Period (PHASE2); Safety-evaluable population (SE)

| | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|
| Treatment duration (days) | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x | xx.x |
| Min-max | xx-xx | xx-xx | xx-xx |
| Treatment duration (days) | | | |

| n | nnn | nnn | nnn |
|------------------------------|-------------|-------------|-------------|
| 1-28 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 29-56 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 57-84 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 85-112 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 113-140 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 141-168 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 169-196 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 197-224 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 225-252 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 253-280 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 281-308 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 309-336 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >= 337 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total cumulative dose (unit) | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X |

| Min-max | xx-xx | xx-xx | XX-XX |
|-----------------------------|-------------|-------------|-------------|
| Number of doses received | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x | xx.x |
| Min-max | xx-xx | xx-xx | xx-xx |
| Number of missed doses | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | XX.X | xx.x |
| Min-max | xx-xx | xx-xx | xx-xx |
| Relative dose intensity (%) | | | |
| n | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x | xx.x |
| Min-max | xx-xx | xx-xx | xx-xx |

# Output 4.2 Concomitant Medications by Medication Class and Preferred Name (CMT01A)

Protocol: GB41149

Analysis Population: Safety-evaluable population

| ATC Class Level 2<br>Other Treatment | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N=nnn) |
|---|---|---|---|
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn | nnn |
| AGENTS ACTING ON THE RENIN-<br>ANGIOTENSIN SYSTEM | | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn | nnn |
| RAMIPRIL | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Class 2 | | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn | nnn |
| Other treatment 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### Output 4.3 Concomitant Medications by Preferred Name (CMT02\_PT)

Protocol: GB41149

Analysis Population: Safety-evaluable population

| Other Treatment | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N=nnn) |
|---|---|---|---|
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn | nnn |
| Other treatment 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Other treatment 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### **Output 4.4 Overview of Deaths and Adverse Events (AET01)**

Protocol: GB41149 Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

| | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|
| Total number of patients with at least one AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of AEs | nn | nn | nn |
| Total number of deaths | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients withdrawn from study due to an AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

| Total number of patients with at least one | | | |
|---|---|---|---|
| AE with fatal outcome | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Serious AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Serious AE leading to withdrawal from treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Serious AE leading to dose modification/interruption | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Related Serious AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| AE leading to withdrawal from treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| AE leading to dose modification/<br>interruption | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Related AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Related AE leading to withdrawal from treatment | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Related AE leading to dose modification/interruption | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Grade 3-5 AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### Output 4.5 Deaths (DTHT01)

Protocol: GB41149

Analysis Population: Safety-evaluable population

| | Placebo MTPS9579A Active (N=xx) (N=xx) | | All patients (N=xxx) |
|---|---|---|---|
| Total number of deaths | nn | nn | nn |

| Primary cause of death | nn | nn | nn |
|------------------------|------------|------------|------------|
| N | | | |
| Adverse event | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Progressive disease | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Other | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Percentages for Total Number of Deaths are relative to total N.

All other percentages are relative to n within each module.

#### Output 4.6 Adverse Events Resulting in Death (AET07)

Protocol: GB41149

Analysis Population: Safety-evaluable population

| MedDRA SOC and Preferred Term | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|
| Total number of deaths | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| SOC1 / PT 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| SOC2 / PT 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| SOC3 / PT 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| SOC4 / PT 4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### **Output 4.7 Adverse Events (AET02)**

Protocol: GB41149 Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)
- (3) 3 patients that were administered saline by IV infusion without IP at week18 visit (DEVI)
- (4) Grade 3+ adverse events (GRD3)

| MedDRA System Organ Class<br>MedDRA Preferred Term | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|
| Total number of patients with at least one adverse event | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Overall total number of events | nn | nn | nn |
| SOC 1 | | | |
| Total number of patients with at least one adverse event | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of events | nn | nn | nn |
| PT 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| PT 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| PT 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| PT 4 | | | |

# Output 4.8 Adverse Events Leading to Study Treatment Discontinuation (AET02)

Protocol: GB41149

Analysis Population: 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

[Similar to output 4.7]

#### Output 4.9 Adverse Events Leading to Study Discontinuation (AET02)

Protocol: GB41149

Analysis Population: 48-Week Double-Blind Treatment Period; Safety-evaluable population

[Similar to output 4.7]

### **Output 4.10 Serious Adverse Events (AET02)**

Protocol: GB41149
Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

[Similar to output 4.7]

#### **Output 4.11 Adverse Events Related to Study Treatment (AET09)**

Protocol: GB41149 Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

[Similar to output 4.7]

#### Output 4.12 Serious Adverse Events Related to Study Treatment (AET02)

Protocol: GB41149 Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

[Similar to output 4.7]

### Output 4.13 Adverse Events by Preferred Term (AET02)

Protocol: GB41149
Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1 PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

| | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|
| MedDRA Preferred Term | | | |
| Total number of patients with at least one adverse event | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Overall total number of events | nn | nn | nn |
| PT 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| PT 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| PT 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| PT 4 | | | |

### Output 4.14 Adverse Events by Highest WHO Toxicity Grade (AET04)

Protocol: GB41149 Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

| MedDRA System Organ<br>Class<br>MedDRA Preferred<br>Term | Grade | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|---|
| - Any adverse events - | - Any Grade - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Grade 1-2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
|---|---|---|---|---|
| | 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Grade 3-4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Grade 5 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| BLOOD AND LYMPHATIC<br>SYSTEM DISORDERS | | | | |
| - Overall - | - Any Grade - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Grade 1-2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Grade 3-4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Grade 5 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| NEUTROPENIAS | - Any Grade - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Grade 1-2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

| 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
|-----------|------------|------------|------------|
| 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Grade 3-4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Grade 5 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

# Output 4.15 Adverse Event of Special Interest Summary Table (AET01\_AESI)

Protocol: GB41149 Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

| | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|
| Total number of patients with at least one AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of AEs | nn | nn | nn |
| Total number of patients with at least one AE by worst grade | | | |
| Grade 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Grade 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

| Grade 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
|---|---|---|---|
| Grade 4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients with study drug withdrawn due to AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients with dose modified/interrupted due to AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients with treatment received for AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients with all non-fatal AEs resolved | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients with at least one unresolved or ongoing non-fatal AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients with at least one serious AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Total number of patients with at least one related AE | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

# Output 4.16 Adverse Events by System Organ Class and Preferred Term (AET01\_ADA)

Protocol: GB41149 Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1\_PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

| MedDRA System Organ Class MedDRA Preferred Term | ADA-<br>(N = XXX) | ADA+<br>(N = XXX) |
|---|---|---|
| Total number of patients with at least one adverse event | nn (xx.x%) | nn (xx.x%) |
| Overall total number of events | nn | nn |
| SOC 1 | | |
| Total number of patients with at least one adverse event | nn (xx.x%) | nn (xx.x%) |
| Total number of events | nn | nn |
| PT 1 | nn (xx.x%) | nn (xx.x%) |
| PT 2 | nn (xx.x%) | nn (xx.x%) |
| PT 3 | nn (xx.x%) | nn (xx.x%) |
| PT 4 | nn (xx.x%) | nn (xx.x%) |

#### Programming notes:

ADA Evaluable Patients are defined as patients with non-missing ADA status (Either Positive or Negative), ADA status is in the ADAB dataset provided by the MSA team.

### Output 4.17 Laboratory Tests and Change from Baseline by Visit (LBT01)

Protocol: GB41149

Analysis Population: Safety-evaluable population

| Parameter: | <parameter></parameter> | | | | |
|---|---|---|---|---|---|
| Visit | | | Placebo<br>(N = XXX) | MTPS9579A Active<br>(N = XXX) | All Patients<br>(N = XXX) |
| Baseline | Value at Visit | n | XXX | XXX | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) | XXXX (XXX) |
| | | Median | xxxx | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX | XXX - XXXX |
| Day 22 | Value at Visit | n | XXX | xxx | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) | XXXX (XXX) |
| | | Median | xxxx | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX | XXX - XXXX |
| | Change from Baseline | n | XXX | xxx | XXX |
| | | Mean (SD) | XXXX (XXX) | XXXX (XXX) | XXXX (XXX) |
| | | Median | xxxx | XXXX | XXXX |
| | | Min - Max | XXX - XXXX | XXX - XXXX | XXX - XXXX |
| | Percent<br>Change from<br>Baseline | n | xxx | xxx | XXX |
| | | Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| | | Median | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| | | Min - Max | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |

# Output 4.18 Laboratory Test Results with Highest WHO Grade Post-Baseline (LBT07)

Protocol: GB41149

Analysis Population: Double-Blind Treatment Period; Safety-evaluable population (PHASE2\_SE)

| Laboratory Test<br>Direction of Abnormality | Highest<br>WHO Grade | Placebo<br>(N = XXX) | MTPS9579A<br>Active<br>(N = XXX) | All Patients<br>(N = XXX) |
|---|---|---|---|---|
| Absolute neutrophil count | n | nn | nn | nn |
| Low | 1 | nn (xx.x <sup>4</sup> %) | nn (xx.x%) | nn (xx.x%) |
| | 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Any | nn (xx.x <sup>6</sup> %) | nn (xx.x%) | nn (xx.x%) |
| Alkaline phosphatase | n | nn | nn | nn |
| High | 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 3 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | 4 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | Any | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

# Output 4.19 Laboratory Test Results with Highest WHO Grade at Any Time (LBT08)

Protocol: GB41149

Analysis Population: Safety-evaluable population

[Similar to output 4.18]

### Output 4.20 Vital Signs Change from Baseline by Visit (VST01)

Protocol: GB41149

Analysis Population: Safety-evaluable population

<Parameter>

| Placebo | MTPS9579A Active | All Patients |
|---------|------------------|--------------|
| (N=nnn) | (N=nnn) | (N=nnn) |

| Visit | Value at Visit | Change<br>from<br>Baseline | Value at Visit | Change from<br>Baseline | Value at<br>Visit | Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|
| Baseline | | | | | | |
| N | nnn | | nnn | | nnn | |
| Mean (SD) | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) | |
| Median | xx.x | | xx.x | | XX.X | |
| Min-max | XX.X-XX.X | | xx.x-xx.x | | XX.X-XX.X | |
| Day XX | | | | | | |
| n | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | XX.X | xx.x | XX.X | XX.X | XX.X |
| Min-max | XX.X -XX.X | XX.X-XX.X | xx.x-xx.x | XX.X-XX.X | XX.X-XX.X | xx.x-xx.x |
| Day XX | | | | | | |
| n | nnn | nnn | nnn | nnn | nnn | Nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | XX.X | xx.x | XX.X | XX.X | xx.x |
| Min-max | XX.X-XX.X | xx.x-xx.x | XX.X-XX.X | xx.x-xx.x | xx.x-xx.x | XX.X-XX.X |

# Output 4.21 Vital Sign Parameters outside Normal Limits Regardless of Abnormality at Baseline (VST02\_1)

Protocol: GB41149

Analysis Population: Safety-evaluable population

| Assessment | Direction of<br>Abnormality | Placebo<br>(N=nnn) | MTPS9579A Active<br>(N=nnn) | All Patients<br>(N=nnn) |
|---|---|---|---|---|
| Diastolic<br>Blood<br>Pressure | Low | nn/nnn (xx.x%) | nn/nnn (xx.x%) | nn/nnn (xx.x%) |
| | High | nn/nnn (xx.x%) | nn/nnn (xx.x%) | nn/nnn (xx.x%) |

| Systolic<br>Blood<br>Pressure | Low | nn/nnn (xx.x%) | nn/nnn (xx.x%) | nn/nnn (xx.x%) |
|---|---|---|---|---|
| Heart Rate | etc. | nn/nnn (xx.x%) | nn/nnn (xx.x%) | nn/nnn (xx.x%) |
| Temperature | | nn/nnn (xx.x%) | nn/nnn (xx.x%) | nn/nnn (xx.x%) |

# Output 4.22 Vital Sign Parameters outside Normal Limits Among Patients without Abnormality at Baseline (VST02\_2)

Protocol: GB41149

Analysis Population: Safety-evaluable population

[Similar to output 4.21]

#### Output 4.23 ECG Parameters Change from Baseline by Visit (EGT01)

Protocol: GB41149

Analysis Population: Safety-evaluable population

[Similar to output 4.20]

# Output 4.24 ECG Parameters outside Normal Limits Regardless of Abnormality at Baseline (EGT02\_1)

Protocol: GB41149

Analysis Population: Safety-evaluable population

[Similar to output 4.21]

## Output 4.25 ECG Parameters outside Normal Limits Among Patients without Abnormality at Baseline (EGT02\_2)

Protocol: GB41149

Analysis Population: Safety-evaluable population

[Similar to output 4.21]

# Output 4.26 QTcF Actual Values and Change from Baseline by Visit (EGT05\_QTCAT)

Protocol: GB41149

Analysis Population: Safety-evaluable population

| | Placebo | MTPS9579A Active | All Patients |
|--------------------------|------------|------------------|--------------|
| Visit / Category | (N=nnn) | (N=nnn) | (N=nnn) |
| Baseline | | | |
| Value at Visit | | | |
| n | nnn | nnn | nnn |
| <=450 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >450 to <=480 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >480 to <=500 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >500 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Day 22<br>Value at Visit | | | |
| n | nnn | nnn | nnn |
| <=450 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >450 to <=480 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >480 to <=500 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >500 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Change from Baseline | | | |
| n | nnn | nnn | nnn |
| <=30 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >30 to <=60 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| >60 msec | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### Listings

### **Output 4.27 Listing of Drug Administration (EXL01)**

Protocol: GB41149

Analysis Population: Double-Blind Treatment Period; Safety-evaluable population (PHASE2\_SE)

Treatment: xxxx (N=xx)

| Center/<br>Pa ient ID | Visit | Study Day<br>From | Study Day<br>To | y | Treatment | Dose | Unit | Frequenc | cy . | Route |
|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1 | | 1 | 27 | RO12 | 2345678 | 25 | MG | QD | ORAL |
| | Day 28 | | 28 | 55 | RO12 | 2345678 | 25 | MG | QD | ORAL |
| | Day 1 | | 1 | 27 | RO12 | 2345678 | 25 | MG | QD | ORAL |
| | Day 1 | | 1 | 27 | RO12 | 2345678 | 25 | MG | QD | ORAL |
| | Day 28 | | 28 | 55 | RO87 | 7654321 | 50 | MG | QD | ORAL |
| | Day 1 | | 1 | 27 | RO12 | 2345678 | 25 | MG | QD | ORAL |
| | Day 28 | | 28 | 55 | R012 | 2345678 | 25 | MG | QD | ORAL |
| | Day 1 | | 1 | 27 | RO12 | 2345678 | 25 | MG | QD | ORAL |
| | Day 28 | | 28 | 55 | RO12 | 2345678 | 25 | MG | QD | ORAL |

# Output 4.28 Glossary of Concomitant Medication Class, Preferred Name, and Investigator-Specified Terms (CML02A\_GL)

Protocol: GB41149

Analysis Population: Double-Blind Treatment Period; Safety-evaluable population (PHASE2\_SE)

| ATC Class Level 2 | WHODrug Preferred Name | Investigator-Specified Treatment Term |
|---|---|---|
| Class2 1 | • | |
| | Preferrered Name 1 | Investigator Text 1 |
| | | Investigator Text 2 |
| | Preferrered Name 2 | Investigator Text 1 |
| | | Investigator Text 2 |
| Class2 2 | Preferrered Name 1 | Investigator Text 1 |
| | | Investigator Text 2 |
| | Preferrered Name 2 | Investigator Text 1 |
| | _ | |

Preferrered Name 1

**Investigator Text 1** 

Preferrered Name 2

**Investigator Text 1** 

### **Output 4.29 Listing of Deaths (AEL04)**

Protocol: GB41149

Analysis Population: Safety-evaluable population

Treatment: PLACEBO

| Center/<br>Patient ID | Age/Sex/Race | Date of First Study<br>Drug<br>Administration | Day of Last Study<br>Drug<br>Administration | Day of Death | Cause of Death | Autopsy<br>Performed? |
|---|---|---|---|---|---|---|
| | /F/ | | 12 | 62 | Myocardial infarction | Yes |
| | /M/ | | 36 | 37 | Ischemic Stroke | No |

#### **Output 4.30 Listing of Pregnancy Results**

Protocol: GB41149

Analysis Population: Safety-evaluable population

Treatment: PLACEBO

| Center/Patient ID | Age/Sex/Race | Type of Sample | Visit | Date of Collection | Pregnancy Result Result | Unit |
|---|---|---|---|---|---|---|
| | /F/ | Blood<br>Blood | SCREENING<br>SCREENING | | | mU/mL |
| | | 2.000 | | 10011010 | | |

### Output 4.31 Glossary of Adverse Event Preferred Terms and Investigator-Specified Adverse Event Terms (AEL01\_NOLLT)

Protocol: GB41149

| MedDRA System Organ Class | MedDRA Preferred Term | Investigator-Specified Adverse Event<br>Term |
|---|---|---|
| BLOOD AND LYMPHATIC<br>SYSTEM DISORDERS | | |
| | ANAEMIA NOS | ANAEMIA |
| | | ANEMIA |
| | LEUCOCYTOSIS NOS | LEUKOCYTOSIS |
| | LEUCOPENIA NOS | LEUKOPENIA |
| | LYMPHADENOPATHY | NECROTIC LYMPH NODE |
| | | SWOLLEN GLANDS IN THROAT |
| | | SWOLLEN THROAT GLANDS |
| | NEUTROPENIA | NEUTROPENIA |
| CARDIAC DISORDERS | | |
| | CARDIOMYOPATHY NOS | CARDIOMYOPATHY |
| | CONGESTIVE (DILATED)<br>CARDIOMYOPATHY | DILATED CARDIOMYOPATHY |
| | PERICARDIAL HAEMORRHAGE | PROBABLE PERICARDIAL BLEED |
| | TACHYCARDIA NOS | TACHYCARDIA |

#### Output 4.32 Listing of Adverse Events (AEL02\_ED)

Protocol: GB41149
Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1 PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2 SE)
- (3) 3 patients that were administered saline by IV infusion without IP at week18 visit (DEVI)

Treatment: <Treatment>

| Center/Patient ID<br>Adverse Event<br>MedDRA<br>Preferred Term | Age/Sex/Race | Study Day<br>at Onset | Time from<br>Last Dose<br>to Onset<br>days hrs mins | AE<br>Duration<br>in Days | Serious | Most<br>Extreme<br>Intensity | Cause<br>d by<br>Study<br>Drug | Outcome (1) | Treatment<br>for AE | Action<br>Taken<br>(2) |
|---|---|---|---|---|---|---|---|---|---|---|
| | /F/ | | | | | | | | | |
| ANEAMIA NOS | | xxx* | xxx xx xx | 1** | No | Mild | Yes | 2 | No | 2 |
| APPETITE DECR | EASED | xxx | xxx xx xx | 2 | No | Moderate | No | 3 | No | 3 |
| | /M <i>i</i> | | | | | | | | | |
| DIARRHEA NOS | | xxx | xxx xx xx | 2** | No | Mild | No | 3 | No | 2 |

<sup>(1)</sup> Outcome: 1 = fatal; 2 = not recovered/not resolved; 3 = recovered/resolved; 4 = recovered/resolved with sequelae; 5 = recovering/resolving; 6 = unknown.

#### **Output 4.33 Listing of Serious Adverse Events (AEL03)**

Protocol: GB41149
Analysis Population:

- (1) Placebo Run-in Period; Run-in safety-evaluable population (PERIOD1 PEFL)
- (2) 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

Treatment: PLACEBO

<sup>(2)</sup> Action taken: 1 = dose increased; 2 = dose not changed; 3 = dose reduced; 4 = drug interrupted; 5 = drug withdrawn; 6 = not applicable; 7 = unknown.

<sup>\*</sup> Study day derived from imputed onset date

<sup>\*\*</sup> Duration derived from imputed onset date and/or end date

| Center/Patient ID<br>SAE MedDRA<br>Preferred Term | Age/Sex/Race | Date of First<br>Study Drug<br>Administratio<br>n | Study Day<br>of Onset | AE<br>Duration in<br>Days | Most<br>Extreme<br>Intensity | Caused<br>by<br>Study<br>Drug | Outcom<br>e<br>(1) | Treatment<br>for SAE | Action<br>Taken<br>(2) | Reason<br>Classified<br>as Serious<br>(3) |
|---|---|---|---|---|---|---|---|---|---|---|
| | /F/ | | | | | | | | | |
| ANEAMIA NOS | | | 60* | 1** | Mild | Yes | 2 | No | 2 | 2 |
| APPETITE DECF | REASED | | 91 | 2** | Moderate | No | 3 | No | 3 | 3 |
| | /M | | | | | | | | | |
| DIARRHEA NOS | | | 425 | 2 | Mild | No | 3 | No | 2 | 6 |

<sup>(1)</sup> Outcome: 1 = fatal; 2 = not recovered/not resolved; 3 = recovered/resolved; 4 = recovered/resolved with sequelae; 5 = recovering/resolving; 6 = unknown.

# Output 4.34 Listing of Adverse Events Leading to Study Treatment Discontinuation (AEL02\_ED)

Protocol: GB41149

Analysis Population: 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

[Similar to output 4.32]

## Output 4.35 Listing of Adverse Events Leading to Study Discontinuation (AEL02\_ED)

Protocol: GB41149

Analysis Population: 48-Week Double-Blind Treatment Period and 12-Week Safety Follow-up Period; Safety-evaluable population (PERIOD2\_SE)

[Similar to output 4.32]

<sup>(2)</sup> Action taken: 1 = dose increased; 2 = dose not changed; 3 = dose reduced; 4 = drug interrupted; 5 = drug withdrawn; 6 = not applicable; 7 = unknown <; Withdrawal = withdrawal from study>.

<sup>(3)</sup> Reason classified as serious: 1 = resulted in death; 2 = life threatening; 3 = required or prolonged in patient hospitalization; 4 = disabling; 5 = a congenital anomaly/birth defect in offspring of study subject; 6 = does not meet any of the above serious criteria, but may jeopardize the subject, and may require medical or surgical intervention to prevent one of the outcomes listed above

<sup>\*</sup> Study day derived from imputed onset date

<sup>\*\*</sup> Duration derived from imputed onset date and/or end date

# Output 4.36 Listing of Laboratory Abnormalities (including WHO grade) (LBL02A)

Protocol: GB41149

Analysis Population: Safety-evaluable population

TREATMENT: <Treatment>

| Lab Test<br>(Unit) | Center /<br>Patient ID | Study<br>Day | Cycle | Date | Days<br>Since<br>Last Dose<br>of Study<br>Drug | Result | Lab<br>Normal<br>Range | WHO<br>Grade |
|---|---|---|---|---|---|---|---|---|
| <lab test=""><br/>(<unit>)</unit></lab> | | | | | | | | |
| | xxxx/xxx | XX | xx | ddMMMYY | xx | xx | XX-XX | xx |
| | xxxx/xxx | xx | xx | ddMMMYY | xx | xx | xx-xx | xx |
| | xxxx/xxx | xx | xx | ddMMMYY | xx | xx | XX-XX | XX |
| | xxxx/xxx | xx | xx | ddMMMYY | xx | xx | XX-XX | xx |
| | xxxx/xxx | XX | XX | ddMMMYY | XX | xx | xx-xx | xx |
| | xxxx/xxx | XX | xx | ddMMMYY | xx | xx | xx-xx | xx |

### **Output 4.37 Listing of Vital Signs (VSL01)**

Protocol: GB41149

Analysis Population: Safety-evaluable population

#### Treatment: <Treatment>

| | Standard<br>Range: | (bea | e Rate<br>ts/min)<br>-100) | R<br>(brea | oiratory<br>tate<br>ths/min)<br>-20) | Pre<br>(m | lic Blood<br>essure<br>mHg)<br>I-130) | Pre<br>(m | olic Blood<br>essure<br>nmHg)<br>i0-80) | | erature<br>(C)<br>5-37.5) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Center / Patient ID<br>Age/Sex/Race<br>Visit/Time Point | Study Day | Result | Change<br>from BL | Result | Change<br>from BL | Result | Change<br>from BL | Result | Change<br>from BL | Result | Change<br>from BL |
| M/<br>Screening<br>Baseline<br>Day 1/ 1HR | XX<br>XX<br>XX | xx<br>xx/L<br>xx/L | xx | xx<br>xx<br>xx | xx | xx<br>xx<br>xx | xx | xx<br>xx<br>xx | xx | xx<br>xx<br>xx | xx |
| Day 1/ 2HR<br>Day 2/ 24HR<br>xxxxx/xx | xx<br>xx<br>xx | xx<br>xx<br>xx | xx | | | | | | | | |
| xx/xx/xxxxx | | | | | | | | | | | |
| xxxxx/xxx | xx<br>xx | xx<br>xx/H | xx | XX | xx | XX | xx | XX | xx | XX | XX |
| | xx<br>xx | xx / H<br>xx | XX<br>XX | | | | | | | | |

Baseline is the patient's last observation prior to initiation of study drug. Abnormalities are flagged as high (H) or low (L) if outside the Roche standard reference range.

### Output 4.38 Listing of ECG Data (EGL01)

Protocol: GB41149

Analysis Population: Safety-evaluable population

[Similar to output 4.37]

### Section 5. Biomarker (PD) Analysis

The analyses of all PD endpoints will be based on the safety-evaluable population.

#### **Tables**

Below 3 tables will be covered in the Safety Section: Output 4.17 Laboratory Tests and Change from Baseline by Visit (LBT01). So there is no need to duplicate those tables.

- 1. Nasosorption Results and Change from Baseline by Visit and Tests
- 2. Urea-normalized Nasosorption Results and Change from Baseline by Visit and Tests
- 3. Serum Results and Change from Baseline by Visit and Tests

#### Graphs

#### **Output 5.1 Mean Value of Active Tryptase Over Time in Nasosorption**

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO\_SE)

#### Output 5.2 Mean Value of Total Tryptase Over Time in Nasosorption

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO\_SE)

### Output 5.3 Mean Value of Active Tryptase Over Time in Nasosorption - Urea Normalized

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO SE)

### Output 5.4 Mean Value of Total Tryptase Over Time in Nasosorption - Urea Normalized

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO\_SE)

#### Output 5.5 Mean Value of Total Tryptase Over Time in Serum

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (SERUM SE)

### Output 5.6 Mean Percent Change From Baseline of Total Tryptase Over Time in Serum

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (SERUM\_SE)

### Output 5.7 Mean Percent Change From Baseline of Active Tryptase Over Time in Nasosorption

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO SE)

## Output 5.8 Mean Percent Change From Baseline of Total Tryptase Over Time in Nasosorption

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO SE)

## Output 5.9 Mean Percent Change From Baseline of Active Tryptase Over Time in Nasosorption - Urea Normalized

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO SE)

## Output 5.10 Mean Percent Change From Baseline of Total Tryptase Over Time in Nasosorption - Urea Normalized

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO SE)

#### **Output 5.11 Mean Value of Urea Over Time in Nasosorption**

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (NASO\_SE)

#### **Output 5.12 Mean Value of Urea Over Time in Serum**

Protocol: GB41149

Analysis Population: Safety-evaluable population; Nasosorption results (SERUM\_SE)